CLINICAL TRIAL: NCT05047861
Title: Evaluation of Implant Placement in Preserved Socket Using Socket Shield Technique With Autogenous Dentin Graft Versus Preserved Socket Using Socket Shield With Alloplast (Controlled Clinical and Radiographic Study)
Brief Title: Implant Placement in the Preserved Socket Using Socket Shield Technique With Autogenous Dentin Graft Versus Preserved Socket Using Socket Shield With Alloplast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Socket shield_2020
Record Dates: First submitted 2021-09-06; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Teeth Extraction; Tooth Socket
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): patients will receive the implant in the previously preserved socket using Socket shield technique with Alloplastic graft material
  Interventions: Procedure: socket shield technique with autogenous dentin graft
- Control group (Active Comparator): patients will receive the implant in the previously preserved socket shield with Autogenous dentin graft
  Interventions: Procedure: socket shield technique with alloplast graft

INTERVENTIONS:
Procedure: socket shield technique with autogenous dentin graft — The crown of the hopeless tooth will be decoronated with a chamfer diamond bur and a large-head round diamond bur under copious irrigation, until the bone crest level.
  The root will then be sectioned along the long axis into buccal and palatal halves with a long shank fissure bur.
  The lingual root fragment will be carefully retrieved using microperiotome. The remaining buccal root fragment will be thinned and concaved slightly with a long shank fissure bur. The thickness of the buccal root fragment should be at least 1.5 mm to ensure resistance to fracture and resorption.
  The coronal part of this shield will be beveled to make a lingual slope for a better emergence profile with a large head round diamond bur.
  The socket shield will be checked for immobility so the implant could be inserted palatally into the socket shield.
  After the final preparation of the socket shield, Graft will be placed using autogenous dentin graft from the discarded palatal part of the tooth
  Arms: Study group
Procedure: socket shield technique with alloplast graft — The crown of the hopeless tooth will be decoronated with a chamfer diamond bur and a large-head round diamond bur under copious irrigation, until the bone crest level.
  The root will then be sectioned along the long axis into buccal and palatal halves with a long shank fissure bur.
  The lingual root fragment will be carefully retrieved using microperiotome. The remaining buccal root fragment will be thinned and concaved slightly with a long shank fissure bur. The thickness of the buccal root fragment should be at least 1.5 mm to ensure resistance to fracture and resorption.
  The coronal part of this shield will be beveled to make a lingual slope for a better emergence profile with a large head round diamond bur.
  The socket shield will be checked for immobility so the implant could be inserted palatally into the socket shield.
  After final preparation of socket shield, Graft will be placed Alloplast graft
  Arms: Control group

SUMMARY:
Alveolar bone resorption and labial bone plate reduction follow teeth extraction due to the deficiency of blood supply, derived from the loss of periodontal ligaments, and hence the socket shield technique with Bone graft was introduced to preserve the periodontal ligaments related perfusion and preserve socket dimensions for new bone formation.

This study aims to compare implants placed in two differently preserved sockets, the first one preserved using Socket Shield technique with Autogenous Dentin Graft while the other socket preserved using socket shield technique with Alloplastic bone graft material

ELIGIBILITY:
Inclusion Criteria:

* One or more of non-restorable (fractured or decayed) tooth/teeth in the upper aesthetic regions (incisors, premolars).
* Intact labial/buccal periodontal tissues.
* Sufficient bone volume to allow placement of an implant.
* Non-Smoker
* Ability to read and sign an informed consent form

Exclusion Criteria:

* A medical history that contraindicates oral surgical treatment (uncontrolled/untreated diabetes mellitus, immunocompromised status,current radio/chemotherapy of the oral and maxillofacial region, treatment with oral and/or intravenous amino-bisphosponates).
* Untreated periodontal disease. [15,18]
* Vertical root fractures on the buccal aspect. [26]
* Tooth /teeth with horizontal fractures below bone level. [26]
* Tooth /teeth with external or internal resorptions.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in implant stability | immeditely and at 3 months
  it will be measured using Osstell ISQ, or Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant.
  High stability means >70 ISQ, between 60-69 is medium stability and < 60 ISQ is considered as low stability.
change in bone density | at baseline and 3 months
  it will be measured using CBCT
change in bone height | at baseline and 3 months
  it will be measured using CBCT
change in Labio/Bucco-Palatal width | at baseline and 3 months
  it will be measured using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt